CLINICAL TRIAL: NCT06603740
Title: Randomized Study Evaluating Cost of Arthrex Nano Arthroscopy Products in Arthroscopic Knee Meniscectomy Versus Conventional Arthroscopy
Brief Title: Nanoscope Cost Analysis Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AIRR-0211
Record Dates: First submitted 2024-08-21; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Meniscal Tear

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Partial meniscectomy using the Arthrex Nanoscope (Experimental)
  Interventions: Device: Arthrex Nanoscope
- Partial meniscectomy using conventional arthroscopy equipment (Other)
  Interventions: Device: Conventional Arthroscopy without Arthrex Nanoscope

INTERVENTIONS:
Device: Arthrex Nanoscope — Arthrex's all-in-one disposable, 2 mm, chip-on-tip camera system now allows surgeons to miniaturize their treatment solutions
  Arms: Partial meniscectomy using the Arthrex Nanoscope
Device: Conventional Arthroscopy without Arthrex Nanoscope — partial meniscectomy using conventional arthroscopy
  Arms: Partial meniscectomy using conventional arthroscopy equipment

SUMMARY:
The study is a pilot study designed to generate preliminary data regarding the cost of partial meniscectomy using NanoScope versus conventional arthroscopy in a traditional operating room (OR) setting

ELIGIBILITY:
Inclusion Criteria:

1. Subject requires simple partial posterior or mid-body meniscectomy.
2. Subject is 18 - 60 years of age.
3. Subject body mass index (BMI) is 35 or lower (BMI ≤ 35).
4. Subject signed informed consent and is willing and able to comply with all study requirements and follow-up visits.
5. Confirmed meniscal injury by physical exam as per standard of care.
6. Normal mechanical alignment; < 5° varus and < 7° valgus, of the affected knee by clinical assessment or X-Rays as per standard of care

Exclusion Criteria:

1. Subject requires complex repair or anterior meniscectomy.
2. Subject has a concomitant chondral lesion of the ipsilateral knee in addition to meniscal tear.
3. Current bilateral knee injury.
4. Insufficient quantity or quality of bone.
5. Blood supply limitations and previous infections which may retard healing.
6. Congenital ligamentous hypermobility defined by Beighton score 4 or 5.
7. Locked knee or haemarthrosis.
8. Subjects that are skeletally immature.
9. Advanced Osteoarthritis; Kellgren Lawrence ≥ 2
10. Fracture of the lower extremities within 6 months prior to screening.
11. Previous surgery on the affected knee within 12 months prior to screening.
12. Sensitivity to silicone, polyester, nylon, FD&C Blue No. 2 dye and beeswax.
13. Other concomitant disease that would interfere with study outcomes.
14. Subject is included in a vulnerable population (child, prisoner, etc).
15. Conditions that tend to limit the patient's ability or willingness to restrict activities, follow directions, or perform online subject assessments during the healing period.
16. Subject is requesting or receiving Worker's compensation related to the knee injury. -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cost Comparison (TDBC) | Operative Visit
  Cost comparison using the time-drive activity-based costing (TDABC) study design between NanoScope versus conventional arthroscopy for partial meniscectomy in a traditional OR setting.

SECONDARY OUTCOMES:
International Knee Documentation Committee (IKDC) Score | Pre Operative, 2 weeks and 6 weeks post op
  The IKDC Questionnaire is a subjective scale that provides patients with an overall function score. The questionnaire looks at 3 categories: symptoms, sports activity, and knee function. The symptoms subscale helps to evaluate things such as pain, stiffness, swelling and giving-way of the knee.
  The questions prompt an answer 0-10.
  The total score is interpreted as a measure of function with higher scores representing higher levels of function.
Visual Analogue Scale (VAS) | Pre Operative, 2 weeks and 6 weeks post op
  The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. A patient marks a point on the line that matches the amount of pain he or she feels.v

OTHER OUTCOMES:
Knee Injury and Osteoarthritis outcome Score (KOOS) | Pre Operative, 2 weeks and 6 weeks post op
  KOOS is a five-subscale patient-reported instrument intended for use from the time of knee injury to the development of osteoarthritis.
  Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic scales and generic measures
PROMIS Pain Interference 6a scale | preop, 2 weeks post op, and 6 weeks post op
PROMIS Pain Intensity 3a scale | preop, 2 weeks post op, and 6 weeks post op
PROMIS Physical Function 13a scale | preop, 2 weeks post op, and 6 weeks post op

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopedic Rhode Island, Warwick, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No